CLINICAL TRIAL: NCT00352586
Title: Psychopharmacology Investigations of Fear Conditioning in Humans
Brief Title: Effect of D-cycloserine on Extinction of Fear Conditioning
Status: Completed | Type: Observational
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020157; 02-M-0157
Record Dates: First submitted 2006-07-13; First posted 2006-07-14 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-02-01

CONDITIONS: Fear
Keywords: Classical Conditioning; Learning; NMDA; Startle; Eyeblink; Anxiety; Fear Conditioning; Fear Potentiated Startle; Extinction; D-cycloserine; Healthy Volunteer; HV; Normal Control
MeSH Terms: conditions — Anxiety Disorders

SUMMARY:
This study will evaluate whether the drug D-cycloserine (DCS) can improve a type of learning called classical conditioning, in which the brain learns to associate neutral stimuli with stimuli that elicit emotional or physiological responses. DCS is an antibiotic that was initially approved to treat tuberculosis and has been tested in clinical trials over the last decade for enhancing cognitive function. This protocol includes both a pilot study and a main study. The main study will begin after the pilot study ends.

Healthy normal volunteers between 18 and 45 years of age may be eligible for these studies. Candidates will be screened with a medical and psychiatric history and a physical examination that includes blood and urine samples, an electrocardiogram (EKG), hearing test and startle test. The startle test involves recording eyeblink responses to loud noises.

After the screening visit, those enrolled will participate in the pilot or main study, in which their reactions to two types of stimuli-an unpleasant, but harmless, shock to the arm and a mild puff of air to the eye-will be measured and recorded.

- Pilot Study

Session 1 - Participants will receive very brief electric shocks delivered through two electrodes attached to the forearm or fingers and will hear brief loud sounds that may startle. Geometric shapes will be presented on a computer monitor.

Sessions 2 and 3 - The procedure is the same as in session 1, except participants will also be subjected to brief low-intensity tones and airpuffs to the eye.

- Main Study

Participants will undergo the same procedures described in the pilot study, with the following additions:

* They will have an intravenous tube placed in a vein for collecting blood during the test.
* They will take a pill each test day that contains either 100 mg DCS, 500 mg DCS, or a placebo (inactive substance). Subjects assigned to receive DCS will get the active drug on only one of the three test sessions and will be given placebo the other two sessions. The placebo group will receive placebo all three sessions.

In both the pilot and main study, subjects' physiological responses to the stimuli will be recorded. Electrodes will be placed on two fingers (to measure sweat, or electrodermal activity), on the ribcage midway between the waist and armpit (to measure heart rate), and under one eye (to measure eye blink). Pulse will be recorded with a device attached to a finger, and breathing rate will be recorded with a special belt placed around the chest. At various times during the sessions, subjects will fill out questionnaires about their experience. Participants may withdraw from the study at any point.

DETAILED DESCRIPTION:
This protocol examines the effect of two drugs on fear conditioning. Study 1 tests assess whether D-cycloserine (DCS) facilitates extinction of fear conditioning and acquisition of eyeblink conditioning. Study 2 examines whether the calcium channel blocker nimodipine blocks acquisition of fear conditioning and eyeblink conditioning.

Study 1: The demonstration that activation of NMDA receptors is necessary for long-term potentiation suggests that this subclass of amino acid may be involved in certain types of learning and memory. The present project will examine the effect DCS, a partial agonist at the glycine modulatory site on the NMDA receptor, on two associative learning tasks, extinction of fear conditioning and acquisition of eyeblink conditioning. The inability to extinguish intense fear memories is a significant clinical problem. Finding procedures or treatments that facilitate extinction of fear memories is of paramount importance. In animals, extinction of conditioned fear involves an active learning process that is blocked by NMDA antagonists. Recently, Dr. Michael Davis (Emory University) demonstrated that the administration of DCS prior to extinction produces a dose-dependent facilitation of extinction of conditioned fear in the rat, when assessed with fear-potentiated startle. We propose to examine whether the clinically important process of extinction can also be enhanced by DCS in humans. Another aim of the study is to examine whether DCS facilitates a hippocampal-mediated task, trace eyeblink conditioning. The hippocampus is particularly rich in NMDA receptors and DCS blocks trace eyeblink conditioning in the rabbit. The present study will examine the effect of placebo, 100 mg DCS, and 500 mg DCS on extinction, retention, and reinstatement of fear-potentiated startle conditioning and acquisition of trace eyeblink conditioning. The first experimental session (acquisition) will be a fear conditioning procedure (paired presentation of a conditioned stimulus or CS and a mildly unpleasant shock). During the second experimental session (extinction), DCS or placebo will be given to the subjects 1 hour prior to an extinction procedure (CS presented without shock). Following extinction, the eyeblink conditioning study will be conducted. Finally, in the third experimental session, retention of fear and eyeblink conditioning will be evaluated. We hypothesized that compared to placebo, DCS will speed up learning, i.e., it will facilitate extinction of fear conditioning and acquisition of eyeblink conditioning.

Study 2: The rationale for testing nimodipine is highly similar to the rationale for testing DCS, and the procedure is very similar. Understanding the neurochemical bases of fear acquisition and fear extinction may provide insights into pathological anxiety and help develop more effective treatments. This study will be conducted over two experimental sessions (and a screening session). Nimodipine or placebo will be given during the 1st session prior to acquisition of fear conditioning and eyeblink conditioning. The 2nd session will be a test of retention of eyeblink conditioning. We hypothesized that nimodipine will impair fear conditioning and eyeblink conditioning.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects must meet the following inclusion criteria in order to participate in the study:

Male or female volunteers ages 18-50 years old.

Judged to be in good physical health on the basis of medical history and physical examination.

Able to understand procedures and agree to participate in the study by giving written informed consent.

EXCLUSION CRITERIA:

Exclusion criteria will be different for studies with and without (pilot study) DCS. Subjects will be excluded from the DCS study if they meet the following exclusion criteria:

* History of allergy to D-cycloserine (study 1) or nimodipine (study 2).
* No clinically significant organ disease by history, physical examination, LFT's, TFT's, electrolytes, BUN, creatinine, Ca+2, Mg+2, urinalysis, CBC with differential, and EKG.
* History of any disease, which in the investigators' opinion may confound the results of the study, including, but not limited to, history of organic mental disorders, seizure, or mental retardation.
* Any significant medical or neurological problems (e.g. cardiovascular illness, respiratory illness, neurologic illness, seizure, stroke, multiple sclerosis, Alzeimer's disease, etc.)
* Past or current substance dependence.
* Presence of psychotropic medications or illicit substance in urine.
* Positive pregnancy test.
* Current or past Axis I psychiatric disorders as identified with the Structured Clinical Interview for DSM-IV-TR axis disorders, non-patient edition (SCID-np).
* Current psychotropic medication.
* Impaired hearing defined as inability to hear a 40 dB(HL) pure tone in the 1000- to 4000 Hz span. Reduced or excessive startle reactivity.
* Neurological symptoms that affect the arms or wrist (e.g., carpal tunnel syndrome).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160
Dates: Start 2002-04-03; Study Completion 2008-02-01

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Gorman JM, Kent JM, Sullivan GM, Coplan JD. Neuroanatomical hypothesis of panic disorder, revised. Am J Psychiatry. 2000 Apr;157(4):493-505. doi: 10.1176/appi.ajp.157.4.493. PMID 10739407